CLINICAL TRIAL: NCT01560169
Title: Clinical Evaluation of Three Celiac Disease-Specific Patient Reported Outcome Instruments in Established and Newly Diagnosed Celiac Disease Patients
Brief Title: Evaluation of Patient Reported Outcome Instruments in Celiac Disease Patients
Status: Completed | Type: Observational
Sponsor: Alvine Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALV003-1121
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Coeliac Disease; Celiac Sprue; Keilakia Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gluten challenge: Gluten containing or gluten-free study food in established celiac disease patients
- Observation: Observation in newly diagnosed celiac disease patients

SUMMARY:
This is an evaluation of celiac-specific patient reported outcome instruments in celiac disease patients.

ELIGIBILITY:
Inclusion Criteria:

* History of biopsy proven celiac disease
* Adherence to a gluten-free diet (established patients only)
* TG2 negative (established patients only)
* TG2 positive (newly diagnosed patients only)
* Signed informed consent

Exclusion Criteria:

* History of IgE-mediated reactions to gluten
* Significant laboratory abnormalities
* History of untreated or GI disease
* Positive pregnancy test
* Any medical condition which could adversely affect study participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Biopsy proven celiac disease patients
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in symptoms using patient reported outcome instruments | 8 and 12 weeks
  Sensitivity of the patient reported outcome instruments to detect change over time in celiac disease symptoms with and without a gluten challenge

SECONDARY OUTCOMES:
Safety - incidence of adverse events | 8 and 12 weeks
  Safety will be evaluated by incidents of adverse events including clinical significant laboratory evaluations and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Adelman, MD, Study Chair — Alvine Pharmaceuticals Inc.
Locations (10):
- United States (9):
  - University of California, San Diego, La Jolla, California
  - Kaiser Permanente Southern California, Allergy Department, San Diego, California
  - University of Colorado, Denver, Aurora, Colorado
  - University of Chicago Celiac Disease Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- University of Alberta, Edmonton, Alberta, Canada